CLINICAL TRIAL: NCT02953483
Title: Ex Vivo Lung Perfusion : Evaluating the Effect of Cellular Perfusate on Mechanical Properties and Gas Exchange Function of the Donor Lungs : A Randomised Cross Over Study
Brief Title: Ex Vivo Lung Perfusion : Effect of Cellular Perfusate on Mechanical Properties and Gas Exchange Function of Donor Lungs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Rajarajan Ganesan, Senior resident, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 10735-PG-1Trg-15/4913-14
Record Dates: First submitted 2016-10-28; First posted 2016-11-02 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-10

CONDITIONS: Organ Preservation
Keywords: Ex Vivo lung perfusion
MeSH Terms: interventions — Erythrocyte Count

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acellular first (Experimental): Lung preservative solution without red blood cells will be used for perfusion in the initial 2 hours followed by addition of red blood cells for the next two hours
  Interventions: Other: Red blood cells
- Cellular first (Experimental): Lung preservative solution will contain red blood cells for the first two hours followed by acellular perfusate for the next two hours
  Interventions: Other: Red blood cells

INTERVENTIONS:
Other: Red blood cells — Packed red blood cells to final hematocrit of 14%

SUMMARY:
The lungs retrieved from the brain dead multi organ donor will be placed in a lab . They will be connected to a ventilator and preservative solution will be circulated through it . Blood will be added to the fluid depending on the group to which the lungs are allocated and its effects on lung function will be seen

DETAILED DESCRIPTION:
The lungs of a brain dead multi organ donor will be retrieved according to standard protocol. Once a decision is made not to transplant the lungs either because of not satisfying ideal criteria or in the absence of a potential recipient they will be included in the study.They will be ventilated optimally and connected to a cardiopulmonary bypass machine for circulating preservative solution through it . Red blood cells will be added to the solution either initially or later depending on the group to which it is allocated .Monitoring of mechanical and gas exchange function and pathological examination of the lungs will be performed at various time points to observe the effect of red blood cells. The lungs will be properly discarded at the end of the procedure and will not be used for transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Brain death certified multi organ donor
* Absence of ideal lung donor criteria or absence of suitable lung recipient

Exclusion Criteria:

* presence of severe mechanical lung injury on visual inspection or radiography
* Presence of pneumonia
* Positive serology ( Hepatitis B,C and HIV

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Compliance | From beginning of perfusion to 4 hours after that
  Measured from the airway pressure on ventilator

SECONDARY OUTCOMES:
Partial pressure to Inspired oxygen concentration ratio | From beginning of perfusion to 4 hours after that
  Ratio of partial pressure of oxygen in perfusate to fraction of inspired oxygen
Pulmonary vascular resistance | From beginning of perfusion to 4 hours after that
  Calculated from measured pulmonary artery pressure and pump flow
Lung injury score | From beginning of perfusion to 4 hours after that
  By pathological examination

CONTACTS AND LOCATIONS:
Overall Officials: Goverdhan D Puri, MD, PhD, Study Director — Post Graduate Institute of Medical Education and Research, Chandigarh
Locations (1):
- Postgraduate Institute of Medical Education and Research, Chandigarh, Chandigarh, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cypel M, Yeung JC, Liu M, Anraku M, Chen F, Karolak W, Sato M, Laratta J, Azad S, Madonik M, Chow CW, Chaparro C, Hutcheon M, Singer LG, Slutsky AS, Yasufuku K, de Perrot M, Pierre AF, Waddell TK, Keshavjee S. Normothermic ex vivo lung perfusion in clinical lung transplantation. N Engl J Med. 2011 Apr 14;364(15):1431-40. doi: 10.1056/NEJMoa1014597. PMID 21488765
- [Background] Yeung JC, Cypel M, Machuca TN, Koike T, Cook DJ, Bonato R, Chen M, Sato M, Waddell TK, Liu M, Slutsky AS, Keshavjee S. Physiologic assessment of the ex vivo donor lung for transplantation. J Heart Lung Transplant. 2012 Oct;31(10):1120-6. doi: 10.1016/j.healun.2012.08.016. PMID 22975103